CLINICAL TRIAL: NCT05801757
Title: Sedative Effect of Remidazolam Besylate Continuous Pump Infusion for Colonoscopic Polypectomy in Elderly Patients
Brief Title: Continuous Infusion of Remidazolam for Colonoscopic Polypectomy in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIRC
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Colon Disease
Keywords: colonoscopic polypectomy; elderly patients
MeSH Terms: conditions — Colonic Diseases | interventions — remimazolam; Propofol

STUDY DESIGN:
Intervention Model Description: Single blind, prospective, randomized controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol group (Active Comparator): propofol 2-3mg/kg/h
  Interventions: Drug: Propofol
- R1 group (Experimental): remimazolam 0.5mg/kg/h
  Interventions: Drug: Remimazolam
- R2 group (Experimental): remimazolam 0.75mg/kg/h
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Using two different doses of remidazolam for continuous pumping to maintain anesthetic effect
  Other Names: Remimazolam besylate
  Arms: R1 group; R2 group
Drug: Propofol — propofol 2-3mg/kg/h
  Other Names: Diprivan
  Arms: Propofol group

SUMMARY:
To observe the sedative effect of continuous infusion of remidazolam in elderly patients undergoing colonoscopic polypectomy.

DETAILED DESCRIPTION:
To observe the sedative effect of continuous infusion of remidazolam in elderly patients undergoing colonoscopic polypectomy, and to screen the optimal dose of remidazolam, in order to provide a more reasonable and safe sedative and analgesic drug regimen for elderly outpatients undergoing colonoscopic polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years old;
* ASA Level I - III;
* Operation time: 15min~1h;
* BMI18.0-29.9；

Exclusion Criteria:

* Emergency surgery;
* Patients with high risk of gastric satiety and reflux aspiration;
* Allergies to benzodiazepines and opioids;
* Those who have taken sedative, analgesic, or antidepressant drugs within 24 hours;
* Abnormal liver and kidney function;
* Previous drug use history;
* Recently participated in other clinical studies;
* Patients who cannot cooperate with communication.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Sedation success rate | 1 day
  Evaluating the success rate of sedation using the modified MOAA/S scoring table

SECONDARY OUTCOMES:
Intraoperative time record | Intraoperative
  Anesthesia time; Operation time; Wake up time; PACU time
Drug usage | 1 day
  doses of propofol,remimazolam and other drugs used
The incidence of adverse reactions during surgery | 1 day
  includes: body movements, hypoxemia, hypotension, bradycardia; Intraoperative awareness
Incidence of postoperative adverse reactions | 24 hours after surgery
  Postoperative nausea and vomiting, postoperative pain, hypotension, bradycardia, dizziness

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
You can request it from the main researcher